CLINICAL TRIAL: NCT00502866
Title: The Feasibility of Assessing the Prevalence of Rickets in Children
Brief Title: Study to Assess the Use of a Simple Lab Test to Screen for Rickets in Children
Status: Completed | Type: Observational
Sponsor: Agency for Healthcare Research and Quality (AHRQ) (U.S. Federal Agency)
Collaborators: University of Washington (Other)
Responsible Party: Sponsor
Other Study IDs: R03HS016029-01 (AHRQ); R03HS016029-01 (AHRQ)
Record Dates: First submitted 2007-07-17; First posted 2007-07-18 (Estimated); Last update posted 2014-01-08 (Estimated); Status verified 2006-10

CONDITIONS: Rickets
Keywords: breastfeeding; vitamin D supplementation; rickets
MeSH Terms: conditions — Rickets; Breast Feeding

STUDY DESIGN:
Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- breastfed children: children, 6-15 months old, predominately breastfed for at least 6 months without supplemental vitamin D

SUMMARY:
Some experts recommend that all breastfed babies receive supplemental vitamin D. The purpose of this study is to determine the rate of vitamin D use in breastfed babies, the recommendations of pediatricians regarding vitamin D, and the impact on these recommendations on parental choice of vitamin D. In addition, in preparation for a large study to see how many breastfed children who don't receive supplemental vitamin D have rickets, in this study we will determine if a simple blood test, an alkaline phosphatase level, could be used to screen for rickets. Parents of children 6-23 months old are eligible to complete feeding surveys and children 6-15 months old who were breastfed for at least the first six months of life and didn't routinely receive vitamin D are eligible for alkaline phosphatase levels. We postulate that most breastfed babies don't receive supplemental vitamin D, and that alkaline phosphatase levels will only be abnormal in a few babies who will have evidence on x-ray of rickets.

DETAILED DESCRIPTION:
The Puget Sound Pediatric Research Network (PSPRN) is a practice-based research network of pediatricians in the Puget Sound area and at the University of Washington and Children's Hospital and Regional Medical Center. The network has extensive experience in conducting large studies on contentious issues that are pertinent to children, their parents, and primary care providers. In 2004, vitamin D supplementation was recommended for all exclusively breastfed infants. This recommendation was based on sporadic reports over the last 30 years of vitamin D deficient rickets in infants and toddlers who have been exclusively breastfed. The recommendation has been controversial because it might undermine efforts to promote breastfeeding, and because the prevalence of rickets in these patients is unknown. PSPRN proposes to conduct a preliminary study to determine the feasibility of a larger planned project by the network to determine the prevalence of rickets in breastfed infants and toddlers who do not receive supplemental vitamin D. Systematic surveys will be conducted in PSPRN practices to determine current levels and trends in vitamin D supplementation. Current practices of PSPRN pediatricians regarding supplementation, and their effect on parents, will also be assessed. The utility of a serum alkaline phosphatase level as a screening test for vitamin D deficient rickets will be determined in the proposed study by obtaining levels on approximately 300 patients, 6-15 months old, seen by PSPRN practitioners, who have been breastfed. In addition to assessing possible methodologies for the larger project, the preliminary study is designed to yield standalone results with important implications.

ELIGIBILITY:
Inclusion Criteria:

* Predominantly breastfed for first 6 months of life
* No routine use of vitamin D during first six months of life
* Singleton birth
* Birth at > 35 weeks gestation

Exclusion Criteria:

* Formula fed
* Significant formula supplementation

Ages: 6 Months to 15 Months | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Study Population: breastfed children
Sampling Method: Non-Probability Sample
Enrollment: 246 (Actual)
Dates: Start 2006-06; Study Completion 2008-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: James A Taylor, MD, Principal Investigator — University of Washington
Locations (1):
- University of Washington, Seattle, Washington, United States

REFERENCES:
- [Result] Taylor JA, Richter M, Done S, Feldman KW. The utility of alkaline phosphatase measurement as a screening test for rickets in breast-fed infants and toddlers: a study from the puget sound pediatric research network. Clin Pediatr (Phila). 2010 Dec;49(12):1103-10. doi: 10.1177/0009922810376993. Epub 2010 Aug 19. PMID 20724326